CLINICAL TRIAL: NCT03450681
Title: Efectividad de la Radiofrecuencia Pulsada Del Nervio Safeno en el Manejo Del Dolor en Artroplastia de Rodilla
Brief Title: Effectiveness of Pulsed Radiofrequency of the Saphenous Nerve in the Management of Knee Arthroplasty Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Carlo Guerrero Nope, anesthesiologist specialist in pain management, Fundación Santa Fe de Bogota
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCEI-2214-2014
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Arthroplasty; Replacement; Knee; Pain
Keywords: Pain Management; Knee Replacement Arthroplasty; Postoperative Pain; Pulsed Radiofrequency Treatment
MeSH Terms: conditions — Pain; Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No pulsed radiofrequency (Placebo Comparator): Procedure consists of a mock incision at the pulsed radiofrequency needle insertion site and standard perioperative pain management by the pain clinic (femoral catheter and PCA)
  Interventions: Procedure: Mock incision
- Pulsed Radiofrequency (Experimental): Procedure consists in pre-operative pulsed radiofrequency under ultrasound guidance of the saphenous nerve and standard postoperative pain management by the pain clinic (femoral catheter and PCA)
  Interventions: Procedure: Pulsed radiofrequency of the saphenous nerve before knee replacement surgery

INTERVENTIONS:
Procedure: Pulsed radiofrequency of the saphenous nerve before knee replacement surgery — A trained anesthesiologist and pain clinician performs ultrasound guided pulsed radiofrequency on the saphenous nerve of a patient undergoing knee replacement surgery, prior to the beginning of the surgical act.
  Arms: Pulsed Radiofrequency
Procedure: Mock incision — A trained anesthesiologist and pain clinician performs a mock incision on the pulsed radiofrequency needle insertion site
  Arms: No pulsed radiofrequency

SUMMARY:
Approximately 40% of patients undergoing total knee arthroplasty develop acute to moderate post operative pain. Furthermore 20-30% develop chronic post operative pain. The objective of this work is to study the effectiveness and safety of pulsed radiofrequency of the saphenous nerve realized during the pre-operative period of total knee arthroplasty. The study design is a randomized, blinded clinical trial. Patients scheduled for total knee arthroplasty are divided into two groups. The first group procedure consists in pre-operative pulsed radiofrequency under ultrasound guidance of the saphenous nerve and standard postoperative pain management by the pain clinic. The second group receives only the standard postoperative pain management by the pain clinic. Patient follow ups are performed 3 times (after 2 weeks, 2 months and 6 months) within a period of 6 months, evaluating pain severity using the VAS.

DETAILED DESCRIPTION:
Methods

Study Design

Randomized, blinded clinical trial. Patients are divided into two groups, one to saphenous nerve block with pulsed radiofrequency guided by ultrasound is applied plus standard pain management by the Pain Clinic, the other one only standard pain management by the Pain Clinic. A 6-month follow-up is evaluating pain by VAS and function by the WOMAC scale

Objectif

Asses the effectivity and safety of preoperatory saphenous nerve pulsed radiofrecuency in total knee arthroplasty between 2014 and 2015 in the Fundación Santa Fe de Bogotá Hospital.

Statistical Analysis

Sample size was calculated using "Sample Size 1.0". The following parameters where used to calculate the sample size for a clinical trial:

Two tails, type I error independent variables 5%, type II error 20%, outcome variable: visual analogue scale from 0 to 100 mm, with a standard deviation of 10 mm and a relevant clinical difference between groups of 20 mm. Additionally, the WOMAC scale, from 0 to 96 points, with a standard deviation of 17 and a relevant clinical difference of 20 points between groups for the three subscales: pain, rigidity and functional capacity, normalized to 100 points each.

A sample size of 41 patients per group is calculated. An adjustment of 20% to compensate possible losses is applied, to a total of 50 patients per group.

Once gathered, the data is processed using the statistical program "Wizard" version 1.7.17. posteriorly, variables are standardized and a descriptive analysis is performed.

Central tendency and dispersion measures are performed to the continuous variables. Percentage distribution and proportion measures are calculated to the categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the Center for Care of Articular Replacements from Fundación Santa Fe University Hospital programed for knee replacement surgery.
* ASA I-III
* Informed consent
* Unilateral Knee Replacement

Exclusion Criteria:

* Neurologic conditions associated with hyperalgesia or allodynia
* Cognitive impairment
* Psychiatric conditions
* Contraindication for the use of local anesthetics
* Bleeding disorders
* Pacemaker or ICD
* Septic arthritis or any infection in the surgical site
* Additional surgical procedure during the surgical act

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pain 6 months after sugery | 6 months
  VAS Pain value 6 months after the knee replacement surgery. The Visual Analog Scale to assess pain ranges from 0mm to 100mm, where 0 is the 'absence of pain' and 100 is 'the worst pain imaginable by the patient'. Lower values in the scale represent a better outcome for the patient.

SECONDARY OUTCOMES:
Opioid consumption during the postoperative period | 3 days
  PCA opioid consumption during postoperative days 0 - 3 in morphine equivalents
Pain on postoperative days 0-3 | 3 days
  VAS Pain value on day 0, 1, 2 and 3 after the knee replacement surgery. The Visual Analog Scale to assess pain ranges from 0mm to 100mm, where 0 is the 'absence of pain' and 100 is 'the worst pain imaginable by the patient'. Lower values in the scale represent a better outcome for the patient.
Pain on postoperative week 2 | 15 days
  VAS Pain value on day 15 after the knee replacement surgery. The Visual Analog Scale to assess pain ranges from 0mm to 100mm, where 0 is the 'absence of pain' and 100 is 'the worst pain imaginable by the patient'. Lower values in the scale represent a better outcome for the patient.
Pain on postoperative month 2 | 2 months
  VAS Pain value 2 months after the knee replacement surgery. The Visual Analog Scale to assess pain ranges from 0mm to 100mm, where 0 is the 'absence of pain' and 100 is 'the worst pain imaginable by the patient'. Lower values in the scale represent a better outcome for the patient.